CLINICAL TRIAL: NCT02804386
Title: Efficacy and Safety of Zoval (Sofosbuvir) and Ribavirin With or Without Interferon (Hepatitis Eradication Accuracy Trial of Sofosbuvir): An Observational Non-interventional Real Life Trial
Brief Title: Efficacy and Safety of Zoval (Sofosbuvir) and Ribavirin With or Without Interferon
Acronym: HEATS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PharmEvo Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PE/ZOVAL/2016/08
Record Dates: First submitted 2016-06-07; First posted 2016-06-17 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C, Chronic
Keywords: HCV; safety; efficacy; EVR; SVR
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): Sofosbuvir, 400 mg OD for 6 months
  Interventions: Drug: Sofosbuvir

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir (formerly known as GS-7977) is a direct-acting nucleotide polymerase inhibitor that is being developed as an oral drug for the treatment of chronic HCV infection
  Other Names: Zoval

SUMMARY:
Title Efficacy and Safety of Zoval (Sofosbuvir) and Ribavirin with or without Interferon among Pakistani Population: A real life trial Hepatitis Eradication Accuracy Trial of Sofosbuvir (HEATS) Study Design Endpoint Classification: Safety/Efficacy Study Intervention Model: Treatment agents (non-interventional observational study): Real life clinical practice study Masking: Open Label Primary Purpose: Treatment Duration Around 12 Months Study Centre Multi centric Study

DETAILED DESCRIPTION:
Indication Chronic Hepatitis C Virus (HCV) infection (serum HCV RNA level, >10,000 IU per milliliter) with or without cirrhosis Primary Objective o Proportion of participants with sustained virologic response 12/24 weeks after discontinuation of therapy (SVR 12 or 24 weeks) [ Time Frame: Post-treatment Week 12/24 ] [ Designated as safety issue: No ]

SVR 12/24 is defined as HCV RNA < the lower limit of quantification (LLOQ; ie, < 15 IU/mL) 12/24 weeks following the last dose of study medication.

Secondary Objective o Proportion of participants experiencing viral breakthrough [ Time Frame: Up to 12 or 24 weeks ] [ Designated as safety issue: No ] Viral breakthrough is defined as HCV RNA ≥ lower limit of quantification (LLOQ) after having previously had HCV RNA < LLOQ while receiving treatment, confirmed with 2 consecutive values (second confirmation value could be post treatment), or last available on-treatment measurement with no subsequent follow-up values.

* Proportion of participants experiencing viral relapse [ Time Frame: Up to Post treatment Week 12 or 24 ] [ Designated as safety issue: No ] Viral relapse is defined as HCV RNA ≥ LLOQ during the post-treatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available post treatment measurement.
* Proportion of participants with Early Virological Response 4 weeks after start of therapy (EVR4) [ Time Frame: Treatment Week 4 ] [ Designated as safety issue: No ]
* SVR 12/24 is defined as HCV RNA < the lower limit of quantification (LLOQ; ie, < 15 IU/mL) 12/24 weeks following the last dose of study medication.Proportion of HCV RNA within 12 or 24 weeks change from baseline in HCV RNA (log10 IU/mL) [ Time Frame: Up to 12 or 24 weeks ] [ Designated as safety issue: No ]
* Proportion of participants experiencing an adverse event (AE) leading to permanent discontinuation of study medication [ Time Frame: Baseline to Week 12 or 24 ] [ Designated as safety issue: No ] Number of Subjects 5000 patients

Dosing - Sofosbuvir 400 mg tablet taken once daily orally

* Ribavirin twice daily orally

  * 1000 mg in patients with body weights <75 kg
  * 1200 mg in those with weights >75 kg
* Interferon for 12 or 24 weeks Drug duration Duration and combination depends upon the discretion of Principal investigator.

Proposed Duration for Genotype:

Inclusion criteria • Men and women, 18 years of age or older,

* Treatment -Naïve and not responded with the previous therapy
* HCV Relapse
* Patient of HCV waiting for transplant, bridge to transplant
* Cirrhosis
* Not previously enrolled in any trial/study of Sofosbuvir Exclusion criteria o Not given informed consent o Pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 years of age or older,
* Treatment -Naïve and not responded with the previous therapy
* Cirrhosis
* Not previously enrolled in any trial of Sofosbuvir

Exclusion Criteria:

* Not given informed consent
* Pregnancy

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Sustained Viralogical response (SVR) | 12 or 24 weeks after discontinuation of therapy
  HCV RNA LLQ < 10 IU/Ml

SECONDARY OUTCOMES:
Viral break through and relapse after discontinuation | Time duration: Up to 12 or 24 weeks
  Viral break through and relapse after discontinuation [Time duration: Up to 12 or 24 weeks]
Level of (Hepatitis C Virus) HCV RNA | within 12 or 24 weeks from baseline
  Level of HCV RNA within 12 or 24 weeks from baseline in HCV RNA (log10 IU/mL) [ Time Frame: Up to 12 or 24 weeks ]

CONTACTS AND LOCATIONS:
Overall Officials: Zahid Azam, FCPS, Principal Investigator — DUHS
Locations (1):
- Ojha, Duhs, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided